CLINICAL TRIAL: NCT04888260
Title: Associations Between Serum Lipids and Mannose Levels in Coronary Artery Disease Among Nondiabetic Patients
Brief Title: Plasma Mannose Associated Parameter Levels in Nondiabetic Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Ramazan Sbirli, Dr., Kafkas University
Other Study IDs: Clinical-4
Record Dates: First submitted 2021-05-07; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Coronary Artery Disease; Hyperlipidemias
MeSH Terms: conditions — Coronary Artery Disease; Hyperlipidemias | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coronary Artery Disease Group: Patients who underwent angiography at the Department of Cardiology and newly diagnosed as coronary artery disease and who weren't on statin treatment were included in the patient group.
  Interventions: Other: Laboratory parameter levels in blood samples
- Control Group: The control group consisted of healthy people with normal coronary arteries angiographically
  Interventions: Other: Laboratory parameter levels in blood samples

INTERVENTIONS:
Other: Laboratory parameter levels in blood samples — Mannose and lipid parameters (triglyceride, LDL, HDL, VLDL) will be analysed in blood samples by using ELISA method.

SUMMARY:
Aims: Nondiabetic patients have been studied to determine whether modest elevations in plasma mannose levels may be associated with a greater incidence of coronary artery disease (CAD).

Methods: The plasma mannose, lipids (triglyceride, LDL, HDL, LDL, VLDL) and LDH levels were successfully will be evaluated with respect to subsequent coronary artery disease using records 120 nondiabetic patients and 120 healthy volunteers. CAD was identified from myocardial infarction and new diagnoses of angina.

The associations between mannose levels and serum lipid parameters will be investigated.

DETAILED DESCRIPTION:
Coronary artery disease (CAD), also known as coronary heart disease (CHD) or ischemic heart disease (IHD), entails a decrease of blood flow to the heart muscle as a result of plaque build-up in the arteries of the heart. CAD are among the world's leading causes of mortality and morbidity, following rapid change and advancement of cardiovascular diagnosis and treatment methods.

The broad range of lipid molecular species in human plasma and their possible role in human health and disease are topics of great interest. Plasma lipidome is now progressively recognized as a potentially important marker of chronic diseases, but the exact degree of its contribution to the interindividual phenotypic variation in family studies is uncertain .

Associative evidence gathered from plasma lipidomic studies promises vital contributions to biomarker research-an important cornerstone of ongoing efforts to prevent chronic disease. The plasma lipidomic profile of humans is associated with various conditions including obesity and disorders of glucose metabolism, hypertension , cardiovascular diseases.

Plasma lipids are solubilized and distributed by associating them with different protein groups. Most free fatty acids and associated structures with carboxyl functional groups interact with albumin, while more complex lipids are transported and distributed using plasma lipoproteins.

Glycerolipids account for a high proportion of total lipids in plasma and include triacylglycerols (TAGs), diacylglycerols (DAGs), and ether-linked glycerolipids. The total plasma concentration of TAGs, allocated between chylomicrons and very-low-density lipoprotein (VLDL), depends on food intake. It is well known that various acquired or secondary risk factors (including genetic determinants, uncontrolled diabetes mellitus, obesity, and sedentary lifestyle) can cause hypertriglyceridemia, a prevalent type of dyslipidemia that is often associated with premature coronary artery disease.

D-mannose, one of the stereoisomers forms, is a structural isomer of D-glucose and commonly found in biological systems, but L-mannose is generally not found in biological systems. Mannose is transported to mammalian cells by hexose transporters primarily by glucose transporters (GLUTs) present in the plasma membrane. Studies demonstrated that plasma mannose levels in human are associated with incident type 2 diabetes mellitus and cardiocascular diseases. On the other hand, molecular mechanism by which the pathway is induced is still unclear. A recent study showed that human plasma lipidome is pleiotropically associated with the cardiovascular risk factors and death.

In mammalian cells, mannose is joined in glycolysis and gluconeogenesis pathways catalyzed by mannose phosphate isomerase. Mannose is a constituent of normal blood plasma and its concentration is generally elevated in diabetes mellitus and chronic glomerulonephritis . However, studies showed that fructose and mannose levels are significantly reduced in obese individuals . Currently, we have reported that elevated baseline mannose in plasma triggered to GLUT4 and Heksokinase-1 (HK1) associated with a progressive risk of CAD with time.

A cytoplasmic enzyme of lactate dehydrogenase (LDH) found in all body cells which transfers a hydride from one molecule to another. LDH catalyzes the reversible conversion of pyruvate to lactate as a unit of Cori cycle. A cardiac marker of LDH is expressed extensively in body cells and a marker of heart failure .

The aims of the study were to determine whether modest elevations in plasma mannose concentrations, and serum lipids [triglyceride, low density lipoprotein (LDL), high density lipoprotein (HDL) and very-low density lipoprotein (VLDL)] may be associated with a greater incidence of CAD among nondiabetic patients. Because hyperglycemia and/or hydrophilicity is associated with additional risk factors for CAD including hypertension, obesity, aging. Additionally, identifying the molecular and biochemical parameters in plasma associated with risk factors for CAD may have strategic importance in the treatment of these diseases.

The patient and control groups will be initially informed about the study and obtained a written consent. Patients who underwent angiography at the Department of Cardiology and newly diagnosed as coronary artery disease and who weren't on statin treatment will be included in the patient group. The control group will be consisted of healthy people with normal coronary arteries angiographically. Patients with chronic renal failure, chronic liver disease, inflammatory disease, diabetes, insulin resistance, major metabolic or endocrine disease will be also excluded. For this purpose, age and sex matched 120 patients and 120 healthy volunteers will be admitted to study.

Blood samples will be collected as described earlier into EDTA and citrate vacutainers.Total cholesterol, high-density lipoprotein and triglycerides will be measured by a commercially available enzymatic colorimetric assay (Roche, Basel,Switzerland). Glucose, creatinine and the other blood profiles will be determined by standard methods.The samples will be centrifuged at 400xg for 10 min to separate the serum.Biochemical parameters will be measured by using an Abbott ARCHITECH c800(Abbott Laboratories, USA) auto analyser and commercial kits. Serum mannose levels will be determined by enzymatic methods using in the ELISA.

Kolmogrov-Smirnov test will be used to determine whether the group was parametrically distributed. Categorical variables were given as numbers and percentages. If the parameters are parametrically distributed, continuous variables will be expressed as mean ± standard deviation; if the parameters are non-parametrically distributed, continuous variables will be expressed as median (IQR). When parametric test assumptions will be provided, the significance test of difference between two means and one-way analysis of variance will be used to compare independent group differences. When parametric test assumptions were not provided, Mann-Whitney U test will be used to compare independent group differences. The relationships between continuous variables will be analyzed using Spearman correlation analysis, chi-square test will be used for analyzing categorical variables. Furthermore, Receiver Operating Characteristic (ROC) curve analysis was used for the discriminant performance serum mannose levels under investigation. In addition, the relationships between continuous variables will be examined by Spearman correlation analysis. P <0.05 will be considered statistically significant in all examinations.

ELIGIBILITY:
For Patient Group Inclusion Criteria To give written informed consent. To underwent angiography at the Pamukkale University Department of Cardiology To be newly diagnosed as coronary artery disease. Not to be on statin treatment.

Exclusion Criteria

* To be on statin treatment. To underwent angiography at the another department or university. Not to be newly diagnosed as coronary artery disease. To have a chronic renal failure, chronic liver disease, inflammatory disease, diabetes, insulin resistance, major metabolic or endocrine disease.

For Control Group;

Inclusion Criteria

To give written informed consent. To underwent angiography at the Pamukkale University Department of Cardiology. To have normal coronary angiography. Not to be on statin treatment.

Exclusion Criteria

* To be on statin treatment. To underwent angiography at the another department or university. To have a chronic renal failure, chronic liver disease, inflammatory disease, diabetes, insulin resistance, major metabolic or endocrine disease.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient and control groups will be initially informed about the study and obtained a written consent. Patients who underwent angiography at the Department of Cardiology and newly diagnosed as coronary artery disease and who weren't on statin treatment will be included in the patient group. The control group will be consisted of healthy people with normal coronary arteries angiographically. Patients with chronic renal failure, chronic liver disease, inflammatory disease, diabetes, insulin resistance, major metabolic or endocrine disease will also be excluded. For this purpose, age and sex matched 120 patients and 120 healthy volunteers will be admitted to study.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Correlations between mannose levels and serum lipid parameters | 16 Months
  This outcome aims to investigate the correlations between mannose levels and serum lipid parameters in patients who have body mass index under than 25 (kg/m^2) and over than 25 kg/m^2.

SECONDARY OUTCOMES:
Correlations between mannose levels and infection parameters (CRP and others). | 6 months
  This outcome aims to investigate the correlations between mannose levels and serum infection parameters(CRP and others) in patients who have body mass index under than 25 (kg/m^2) and over than 25 kg/m^2.
The effect of comorbidites on correlation between the serum mannose levels and serum lipid parameters and serum infecition parameters | 6 months
  This outcome aims to investigate the effect of comorbidites on correlation between the serum mannose levels and serum lipid parameters and serum infecition parameters in patients who have body mass index under than 25 (kg/m^2) and over than 25 kg/m^2 and in patient who have hypertension disease.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Aylin Koseler, Denizli, Outside of the US
  - Ramazan Sabirli, Kars, Outside of the US

IPD SHARING:
Plan to Share IPD: Undecided
Plan is undecided.